CLINICAL TRIAL: NCT01589107
Title: A Randomized Controlled Trial of a Video Decision Making Aid to Obtain Informed Consent in the Surgical Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011-P-001731
Record Dates: First submitted 2012-04-28; First posted 2012-05-01 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Surgery; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): usual care
- Video Arm (Experimental)
  Interventions: Behavioral: video decision aid

INTERVENTIONS:
Behavioral: video decision aid — video decision aid
  Arms: Video Arm

SUMMARY:
To demonstrate that clinical surrogates of SICU patients who view a video decision aid in addition to receiving written and verbal information about procedures and life sustaining therapy in the SICU make more informed decisions than patients and clinical surrogates who receive written and verbal information alone.

DETAILED DESCRIPTION:
Specific Aim 1: To demonstrate that clinical surrogates of SICU patients who view a video decision aid in addition to receiving written and verbal information about procedures and life sustaining therapy in the SICU make more informed decisions than patients and clinical surrogates who receive written and verbal information alone.

Hypothesis 1: Adding a video decision aid to the current informed consent process, for procedures and life sustaining treatments in the SICU, will better inform clinical surrogates of incapacitated patients admitted to the SICU regarding decision making when providing consent for medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical surrogates of the following patients will be eligible to participate in this opinion survey:

  1. All patients admitted to the SICU and not expected to die within 48 hours.
  2. Patient has been admitted to the acute care surgical service,
  3. The patient is over the age of 50 and does not have decision making capacity.
* Subjects must be over the age of 21 and English speaking to participate in the opinion survey.

Exclusion Criteria:

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
knowledge of risks and benefits of procedures | 5 minutes after survey
  knowledge of risks and benefits of procedures

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Volandes, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States